CLINICAL TRIAL: NCT00000575
Title: Childhood Asthma Management Program
Brief Title: Childhood Asthma Management Program (CAMP) Phases I (Trial), II (CAMPCS), III (CAMPCS/2), and IV (CAMPCS/3)
Acronym: CAMP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); CAMP Steering Committee (Unknown)
Responsible Party: Principal Investigator, James Tonascia, Principal Investigator, CAMP Data Coordinating Center, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 213; 5U01HL075417 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Results first posted 2014-04-03 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-02

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases | interventions — Nedocromil; Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 Budesonide (Active Comparator): Budesonide (Pulmicort), two 100 microgram puffs bid + two microgram puffs albuterol (Ventolin) prn
  Interventions: Drug: Budesonide
- 2 Nedocromil (Active Comparator): Nedocromil (Tilade), four 2 mg puffs bid + two 90 microgram puffs albuterol prn
  Interventions: Drug: Nedocromil
- 3 Placebo (Placebo Comparator): Two 100 microgram puffs budesonide placebo bid + two 90 microgram puffs albuterol prn or four 2 mg puffs nedocromil placebo bid + two 90 microgram puffs albuterol prn.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Two 100 Og puffs budesonide placebo bid + two 90 Og puffs albuterol prn OR four 2 mg puffs nedocromil placebo bid + two 90 Og puffs albuterol prn.
  Arms: 3 Placebo
Drug: Nedocromil — Four 2 mg puffs bid + two 90 Og puffs albuterol prn
  Other Names: Tilade
  Arms: 2 Nedocromil
Drug: Budesonide — Two 100 Og puffs bid + two 90 Og puffs albuterol prn.
  Other Names: Pulmicort
  Arms: 1 Budesonide

SUMMARY:
The purpose of this study is to evaluate the long term effects of anti-inflammatory therapy compared to bronchodilator therapy on the course of asthma, particularly on lung function and bronchial hyperresponsiveness, and on physical and psychosocial growth and development.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma is a serious chronic condition, affecting approximately 14 million Americans. People with asthma experience well over 100 million days of restricted activity annually, and costs for asthma care exceed $10 billion a year. Asthma is much more prevalent among children than adults.

Hospitalizations for asthma have been increasing among children. For example, from 1979 to 1987, the hospital discharge rate with asthma as the first-listed diagnosis rose 43 percent among children less than 15 years of age, from 19.8 to 28.4 discharges per 10,000 population.

Death rates for asthma are greater in Blacks than in whites, and the difference is increasing. In 1979, Blacks of both sexes were about twice as likely to die from asthma as whites. Over the past decade this ratio has increased, and by 1987 the asthma death rate was almost three times greater among Blacks than whites. In children, these mortality differences between Blacks and whites are even more striking.

Current knowledge about the epidemiology and natural history of childhood asthma is incomplete, but the relationship between asthma early in life and development of chronic obstructive pulmonary disease (COPD) in adulthood is becoming more apparent. Asthmatic children with persistent and severe asthma symptoms have lower levels of lung function by young adulthood than those with milder disease. Recent longitudinal studies have confirmed a decrease in rate of growth of lung function as measured by FEV1 among symptomatic (primarily wheeze) children compared to asymptomatic children. Among persons who develop COPD, initial level of lung function is the strongest predictor of subsequent rapid decline of ventilatory function.

Thus, less than maximally attained levels of lung function among children with asthma may predispose them to greater than normal decline of lung function later in life. Although the long-term effect of treatment on the course of asthma is not known, the treatment goal of decreasing bronchial hyperresponsiveness and maximizing lung function and growth during childhood may have a beneficial effect on lung health throughout life and prevent progression to irreversible airflow obstruction.

Two classes of medications are currently available for treatment of inflammation--corticosteroids and cromolyn sodium. Inhaled corticosteroids have significantly fewer side effects than systemic administration. Corticosteroids do not inhibit the early asthmatic response, but are effective in suppressing the inflammation and bronchial hyperresponsiveness of the late phase response. Long-term studies of inhaled corticosteroids have shown beneficial effects on lung function as measured by FEV1. However, there has been concern about possible effects of long-term use of inhaled corticosteroids. Although epidemiological studies of the use of inhaled corticosteroids have shown no significant adverse effects, large-scale randomized controlled studies of their effects on children's growth and development are needed.

When CAMP was initiated in the United States, bronchodilator treatment was the most common approach to therapy. Two classes of bronchodilators, inhaled beta-2-adrenergic agonists and oral theophylline, are most frequently prescribed for asthma. To date, no randomized, controlled studies have compared the two classes of anti-inflammatory medications to each other and to bronchodilator therapy on the course of asthma.

The initiative was proposed by the Pulmonary Disease Advisory Committee working group in October 1987 and approved by the full committee at the February 1988 meeting and by the National Heart, Lung, and Blood Advisory Council in May 1990. The Request for Proposals was released in October 1990. Awards were made in September 1991.

DESIGN NARRATIVE:

Children were randomized to one of three treatment groups to receive either: inhaled albuterol alone, albuterol with inhaled budesonide, albuterol with nedocromil. Upon randomization, data were collected on demographic factors, physical and psychosocial development, clinical factors including medical history and extent of allergies, and quality of life factors including limitation of activity, absenteeism from school, emergency room visits, and hospitalizations. All subjects received a common educational program, differing only in the information presented regarding the medication used by the subjects. Each subject was given a standard protocol for dealing with asthma attacks. All subjects were treated and followed for five years with quarterly visits yearly. Recruitment began in July 1993 and ended in June 1995 with the accrual of 1,041 subjects.

The study has been extended through June 2011 through three funding phases to observe the subjects but not provide asthma treatment. This will allow CAMP to (1.) determine the full impact of 4 to 6 years of anti-inflammatory therapy on attaining maximal lung function and final height; (2.) examine the natural history of asthma through age 26; and (3.) define patterns of reduced lung function growth and early decline of lung function in young adults.

ELIGIBILITY:
Inclusion criteria:

* Age 5 to 12 years at time of screening
* Chronic asthma as evidenced by one or more of the following historical findings for at least 6 months during the past year:
* Asthma symptoms at least 2 times per week
* 2 or more usages per week of an inhaled bronchodilator
* Daily asthma medication
* Current asthma symptoms either by diary symptom code of 1 or greater or am or pm PEFR less than 80% of personal best post-bronchodilator value by diary, on 8 or more days during the prn screening period
* Methacholine sensitivity: estimated PC20 FEV1 less than or equal to 12.5 mg/ml
* Consent of guardian and assent of child
* Ability to comply with trial for 5 - 6.5 years

Exclusion criteria:

* Presence of one or more of the following confounding or complicating problems:
* Any other active pulmonary disease
* Any chronic condition presumed to interfere with the successful completion of the project or confound its interpretation
* Pulmonary function testing findings suggesting a ventilatory defect other than asthma, or evidence of existing irreversible lung damage
* Severe chronic sinusitis or nasal polyposis
* Introduction of or a change in allergen immunotherapy within the past month
* Use of more than 4 sprays of nasal steroids daily (only beclomethasone allowed)
* Pregnancy
* Current use of metoclopramide, ranitidine, or cimetidine
* Treatment for gastroesophageal reflux
* Participation in another drug study
* Evidence of severe asthma as indicated by one or more of the following:
* Two or more hospitalizations for asthma in the past year
* Six or more steroid bursts in the past year
* Demonstrated need for continuous use of glucocorticoids, either oral or inhaled
* When off inhaled O2-agonist for more than 4 hrs and theophylline for more than 24 hrs, FEV1 less than 65% predicted
* Intubation for asthma at any time in the past
* Need for 9 or more puffs/day of albuterol for each of 3 consecutive days (excluding preventive use prior to exercise), or nocturnal asthma awakenings more than 1.5 times per week on average, or average diary card symptom code greater than 2, or requirement for other medications to control asthma, during prn screening period
* Inability to perform 3 acceptable FVC maneuvers of which at least 2 reproducible FEV1s are within 10% of the largest FEV1
* Inability to complete the methacholine challenge or methacholine PC20 FEV1 greater than 12.5 mg/ml
* Evidence that patient or family may be unreliable or non-compliant or may move from the metropolitan area before trial completion

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1041 (Actual)
Dates: Start 1991-09; Primary Completion 1999-10 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: N. F. Adkinson, MD, Principal Investigator — Johns Hopkins University; Anne Fuhlbrigge, MD, MS, Principal Investigator — Brigham and Women's Hospital; H. W. Kelly, PharmD, Principal Investigator — University of New Mexico; Padmaja Subbarao, MD, MSc, Principal Investigator — The Hospital for Sick Children; Paul Williams, MD, Principal Investigator — Asthma, Inc.; Robert Strunk, MD, Principal Investigator — Washington University School of Medicine; Stanley Szefler, MD, Principal Investigator — National Jewish Health; James Tonascia, PhD, Principal Investigator — Johns Hopkins University; Robert Zeiger, MD, PhD, Principal Investigator — University of California, San Diego

REFERENCES:
- [Background] Design and implementation of a patient education center for the Childhood Asthma Management Program. Childhood Asthma Management Program Research Group. Ann Allergy Asthma Immunol. 1998 Dec;81(6):571-81. PMID 9892029
- [Background] Recruitment of participants in the childhood Asthma Management Program (CAMP). I. Description of methods: Childhood Asthma Management Program Research Group. J Asthma. 1999 May;36(3):217-37. PMID 10350219
- [Background] The Childhood Asthma Management Program (CAMP): design, rationale, and methods. Childhood Asthma Management Program Research Group. Control Clin Trials. 1999 Feb;20(1):91-120. PMID 10027502
- [Background] Zeiger RS, Dawson C, Weiss S. Relationships between duration of asthma and asthma severity among children in the Childhood Asthma Management Program (CAMP). J Allergy Clin Immunol. 1999 Mar;103(3 Pt 1):376-87. doi: 10.1016/s0091-6749(99)70460-4. PMID 10069869
- [Background] Nelson HS, Szefler SJ, Jacobs J, Huss K, Shapiro G, Sternberg AL. The relationships among environmental allergen sensitization, allergen exposure, pulmonary function, and bronchial hyperresponsiveness in the Childhood Asthma Management Program. J Allergy Clin Immunol. 1999 Oct;104(4 Pt 1):775-85. doi: 10.1016/s0091-6749(99)70287-3. PMID 10518821
- [Background] Bender BG, Annett RD, Ikle D, DuHamel TR, Rand C, Strunk RC. Relationship between disease and psychological adaptation in children in the Childhood Asthma Management Program and their families. CAMP Research Group. Arch Pediatr Adolesc Med. 2000 Jul;154(7):706-13. doi: 10.1001/archpedi.154.7.706. PMID 10891023
- [Background] Larsen GL. Focusing on childhood asthma: the childhood asthma management program (CAMP). J Allergy Clin Immunol. 1999 Mar;103(3 Pt 1):371-3. doi: 10.1016/s0091-6749(99)70458-6. No abstract available. PMID 10069867
- [Background] Weiss ST, Van Natta ML, Zeiger RS. Relationship between increased airway responsiveness and asthma severity in the childhood asthma management program. Am J Respir Crit Care Med. 2000 Jul;162(1):50-6. doi: 10.1164/ajrccm.162.1.9811005. PMID 10903219
- [Background] Annett RD, Aylward EH, Lapidus J, Bender BG, DuHamel T. Neurocognitive functioning in children with mild and moderate asthma in the childhood asthma management program. The Childhood Asthma Management Program (CAMP) Research Group. J Allergy Clin Immunol. 2000 Apr;105(4):717-24. doi: 10.1067/mai.2000.105226. PMID 10756221
- [Background] Childhood Asthma Management Program Research Group; Szefler S, Weiss S, Tonascia J, Adkinson NF, Bender B, Cherniack R, Donithan M, Kelly HW, Reisman J, Shapiro GG, Sternberg AL, Strunk R, Taggart V, Van Natta M, Wise R, Wu M, Zeiger R. Long-term effects of budesonide or nedocromil in children with asthma. N Engl J Med. 2000 Oct 12;343(15):1054-63. doi: 10.1056/NEJM200010123431501. PMID 11027739
- [Background] Huss K, Adkinson NF Jr, Eggleston PA, Dawson C, Van Natta ML, Hamilton RG. House dust mite and cockroach exposure are strong risk factors for positive allergy skin test responses in the Childhood Asthma Management Program. J Allergy Clin Immunol. 2001 Jan;107(1):48-54. doi: 10.1067/mai.2001.111146. PMID 11149990
- [Background] Yu O, Sheppard L, Lumley T, Koenig JQ, Shapiro GG. Effects of ambient air pollution on symptoms of asthma in Seattle-area children enrolled in the CAMP study. Environ Health Perspect. 2000 Dec;108(12):1209-14. doi: 10.1289/ehp.001081209. PMID 11133403
- [Background] Annett RD, Bender BG, Lapidus J, Duhamel TR, Lincoln A. Predicting children's quality of life in an asthma clinical trial: what do children's reports tell us? J Pediatr. 2001 Dec;139(6):854-61. doi: 10.1067/mpd.2001.119444. PMID 11743513
- [Background] Weiss ST, Horner A, Shapiro G, Sternberg AL; Childhood Asthma Management Program (CAMP) Research Group. The prevalence of environmental exposure to perceived asthma triggers in children with mild-to-moderate asthma: data from the Childhood Asthma Management Program (CAMP). J Allergy Clin Immunol. 2001 Apr;107(4):634-40. doi: 10.1067/mai.2001.113869. PMID 11295651
- [Background] Strunk RC, Sternberg AL, Bacharier LB, Szefler SJ. Nocturnal awakening caused by asthma in children with mild-to-moderate asthma in the childhood asthma management program. J Allergy Clin Immunol. 2002 Sep;110(3):395-403. doi: 10.1067/mai.2002.127433. PMID 12209085
- [Background] DeMeo DL, Lange C, Silverman EK, Senter JM, Drazen JM, Barth MJ, Laird N, Weiss ST. Univariate and multivariate family-based association analysis of the IL-13 ARG130GLN polymorphism in the Childhood Asthma Management Program. Genet Epidemiol. 2002 Nov;23(4):335-48. doi: 10.1002/gepi.10182. PMID 12432502
- [Background] Strunk RC, Bender B, Young DA, Sagel S, Glynn E, Caesar M, Lawhon C. Predictors of protocol adherence in a pediatric asthma clinical trial. J Allergy Clin Immunol. 2002 Oct;110(4):596-602. doi: 10.1067/mai.2002.128803. PMID 12373267
- [Background] Kelly HW, Strunk RC, Donithan M, Bloomberg GR, McWilliams BC, Szefler S; Childhood Asthma Management Program (CAMP). Growth and bone density in children with mild-moderate asthma: a cross-sectional study in children entering the Childhood Asthma Management Program (CAMP). J Pediatr. 2003 Mar;142(3):286-91. doi: 10.1067/mpd.2003.86. PMID 12640377
- [Background] Bacharier LB, Dawson C, Bloomberg GR, Bender B, Wilson L, Strunk RC; Childhood Asthma Management Program Research Group. Hospitalization for asthma: atopic, pulmonary function, and psychological correlates among participants in the Childhood Asthma Management Program. Pediatrics. 2003 Aug;112(2):e85-92. doi: 10.1542/peds.112.2.e85. PMID 12897312
- [Background] Tantisira KG, Litonjua AA, Weiss ST, Fuhlbrigge AL; Childhood Asthma Management Program Research Group. Association of body mass with pulmonary function in the Childhood Asthma Management Program (CAMP). Thorax. 2003 Dec;58(12):1036-41. doi: 10.1136/thorax.58.12.1036. PMID 14645968
- [Background] Silverman EK, Kwiatkowski DJ, Sylvia JS, Lazarus R, Drazen JM, Lange C, Laird NM, Weiss ST. Family-based association analysis of beta2-adrenergic receptor polymorphisms in the childhood asthma management program. J Allergy Clin Immunol. 2003 Nov;112(5):870-6. doi: 10.1016/s0091-6749(03)02023-2. PMID 14610472
- [Background] Lange C, Lyon H, DeMeo D, Raby B, Silverman EK, Weiss ST. A new powerful non-parametric two-stage approach for testing multiple phenotypes in family-based association studies. Hum Hered. 2003;56(1-3):10-7. doi: 10.1159/000073728. PMID 14614234
- [Background] Slaughter JC, Lumley T, Sheppard L, Koenig JQ, Shapiro GG. Effects of ambient air pollution on symptom severity and medication use in children with asthma. Ann Allergy Asthma Immunol. 2003 Oct;91(4):346-53. doi: 10.1016/S1081-1206(10)61681-X. PMID 14582813
- [Background] Bender BG, Ellison MC, Gleason M, Murphy JR, Sundstrom DA, Szefler SJ. Minimizing attrition in a long-term clinical trial of pediatric asthma. Ann Allergy Asthma Immunol. 2003 Aug;91(2):168-76. doi: 10.1016/S1081-1206(10)62173-4. PMID 12952111
- [Background] Raby BA, Silverman EK, Lazarus R, Lange C, Kwiatkowski DJ, Weiss ST. Chromosome 12q harbors multiple genetic loci related to asthma and asthma-related phenotypes. Hum Mol Genet. 2003 Aug 15;12(16):1973-9. doi: 10.1093/hmg/ddg208. PMID 12913068
- [Background] Lake SL, Lyon H, Tantisira K, Silverman EK, Weiss ST, Laird NM, Schaid DJ. Estimation and tests of haplotype-environment interaction when linkage phase is ambiguous. Hum Hered. 2003;55(1):56-65. doi: 10.1159/000071811. PMID 12890927
- [Background] Bacharier LB, Raissy HH, Wilson L, McWilliams B, Strunk RC, Kelly HW. Long-term effect of budesonide on hypothalamic-pituitary-adrenal axis function in children with mild to moderate asthma. Pediatrics. 2004 Jun;113(6):1693-9. doi: 10.1542/peds.113.6.1693. PMID 15173493
- [Background] Covar RA, Spahn JD, Murphy JR, Szefler SJ; Childhood Asthma Management Program Research Group. Progression of asthma measured by lung function in the childhood asthma management program. Am J Respir Crit Care Med. 2004 Aug 1;170(3):234-41. doi: 10.1164/rccm.200308-1174OC. Epub 2004 Mar 17. PMID 15028558
- [Background] Tantisira KG, Lake S, Silverman ES, Palmer LJ, Lazarus R, Silverman EK, Liggett SB, Gelfand EW, Rosenwasser LJ, Richter B, Israel E, Wechsler M, Gabriel S, Altshuler D, Lander E, Drazen J, Weiss ST. Corticosteroid pharmacogenetics: association of sequence variants in CRHR1 with improved lung function in asthmatics treated with inhaled corticosteroids. Hum Mol Genet. 2004 Jul 1;13(13):1353-9. doi: 10.1093/hmg/ddh149. Epub 2004 May 5. PMID 15128701
- [Background] Lazarus R, Raby BA, Lange C, Silverman EK, Kwiatkowski DJ, Vercelli D, Klimecki WJ, Martinez FD, Weiss ST. TOLL-like receptor 10 genetic variation is associated with asthma in two independent samples. Am J Respir Crit Care Med. 2004 Sep 15;170(6):594-600. doi: 10.1164/rccm.200404-491OC. Epub 2004 Jun 16. PMID 15201134
- [Background] Covar RA, Szefler SJ, Martin RJ, Sundstrom DA, Silkoff PE, Murphy J, Young DA, Spahn JD. Relations between exhaled nitric oxide and measures of disease activity among children with mild-to-moderate asthma. J Pediatr. 2003 May;142(5):469-75. doi: 10.1067/mpd.2003.187. PMID 12756375
- [Background] Covar RA, Spahn JD, Martin RJ, Silkoff PE, Sundstrom DA, Murphy J, Szefler SJ. Safety and application of induced sputum analysis in childhood asthma. J Allergy Clin Immunol. 2004 Sep;114(3):575-82. doi: 10.1016/j.jaci.2004.06.036. PMID 15356559
- [Background] Randolph AG, Lange C, Silverman EK, Lazarus R, Silverman ES, Raby B, Brown A, Ozonoff A, Richter B, Weiss ST. The IL12B gene is associated with asthma. Am J Hum Genet. 2004 Oct;75(4):709-15. doi: 10.1086/424886. Epub 2004 Aug 20. PMID 15322986
- [Background] Randolph AG, Lange C, Silverman EK, Lazarus R, Weiss ST. Extended haplotype in the tumor necrosis factor gene cluster is associated with asthma and asthma-related phenotypes. Am J Respir Crit Care Med. 2005 Sep 15;172(6):687-92. doi: 10.1164/rccm.200501-122OC. Epub 2005 Jun 23. PMID 15976383
- [Background] Annett RD, Stansbury K, Kelly HW, Strunk RC. Association of hypothalamic-pituitary-adrenal axis function with neuropsychological performance in children with mild/moderate asthma. Child Neuropsychol. 2005 Aug;11(4):333-48. doi: 10.1080/09297040490916929. PMID 16051562
- [Background] Raby BA, Hwang ES, Van Steen K, Tantisira K, Peng S, Litonjua A, Lazarus R, Giallourakis C, Rioux JD, Sparrow D, Silverman EK, Glimcher LH, Weiss ST. T-bet polymorphisms are associated with asthma and airway hyperresponsiveness. Am J Respir Crit Care Med. 2006 Jan 1;173(1):64-70. doi: 10.1164/rccm.200503-505OC. Epub 2005 Sep 22. PMID 16179640
- [Background] Raby BA, Van Steen K, Celedon JC, Litonjua AA, Lange C, Weiss ST; CAMP Research Group. Paternal history of asthma and airway responsiveness in children with asthma. Am J Respir Crit Care Med. 2005 Sep 1;172(5):552-8. doi: 10.1164/rccm.200501-010OC. Epub 2005 Jun 3. PMID 15937295
- [Derived] Li J, Hong X, Jiang M, Kho AT, Tiwari A, Wang AL, Chase RP, Celedon JC, Weiss ST, McGeachie MJ, Tantisira KG. A novel piwi-interacting RNA associates with type 2-high asthma phenotypes. J Allergy Clin Immunol. 2024 Mar;153(3):695-704. doi: 10.1016/j.jaci.2023.10.032. Epub 2023 Dec 4. PMID 38056635
- [Derived] Sordillo JE, Lutz SM, Kelly RS, McGeachie MJ, Dahlin A, Tantisira K, Clish C, Lasky-Su J, Wu AC. Plasmalogens Mediate the Effect of Age on Bronchodilator Response in Individuals With Asthma. Front Med (Lausanne). 2020 Feb 14;7:38. doi: 10.3389/fmed.2020.00038. eCollection 2020. PMID 32118022
- [Derived] Wang AL, Gruzieva O, Qiu W, Kebede Merid S, Celedon JC, Raby BA, Soderhall C, DeMeo DL, Weiss ST, Melen E, Tantisira KG. DNA methylation is associated with inhaled corticosteroid response in persistent childhood asthmatics. Clin Exp Allergy. 2019 Sep;49(9):1225-1234. doi: 10.1111/cea.13447. Epub 2019 Aug 15. PMID 31187518
- [Derived] Sordillo JE, McGeachie M, Lutz SM, Lasky-Su J, Tantisira K, Tsai CH, Dahlin A, Kelly R, Wu AC. Longitudinal analysis of bronchodilator response in asthmatics and effect modification of age-related trends by genotype. Pediatr Pulmonol. 2019 Feb;54(2):158-164. doi: 10.1002/ppul.24219. Epub 2018 Dec 25. PMID 30585438
- [Derived] Kho AT, McGeachie MJ, Moore KG, Sylvia JM, Weiss ST, Tantisira KG. Circulating microRNAs and prediction of asthma exacerbation in childhood asthma. Respir Res. 2018 Jun 26;19(1):128. doi: 10.1186/s12931-018-0828-6. PMID 29940952
- [Derived] McGeachie MJ, Clemmer GL, Croteau-Chonka DC, Castaldi PJ, Cho MH, Sordillo JE, Lasky-Su JA, Raby BA, Tantisira KG, Weiss ST. Whole genome prediction and heritability of childhood asthma phenotypes. Immun Inflamm Dis. 2016 Nov 28;4(4):487-496. doi: 10.1002/iid3.133. eCollection 2016 Dec. PMID 27980782
- [Derived] McGeachie MJ, Yates KP, Zhou X, Guo F, Sternberg AL, Van Natta ML, Wise RA, Szefler SJ, Sharma S, Kho AT, Cho MH, Croteau-Chonka DC, Castaldi PJ, Jain G, Sanyal A, Zhan Y, Lajoie BR, Dekker J, Stamatoyannopoulos J, Covar RA, Zeiger RS, Adkinson NF, Williams PV, Kelly HW, Grasemann H, Vonk JM, Koppelman GH, Postma DS, Raby BA, Houston I, Lu Q, Fuhlbrigge AL, Tantisira KG, Silverman EK, Tonascia J, Strunk RC, Weiss ST; CAMP Research Group. Genetics and Genomics of Longitudinal Lung Function Patterns in Individuals with Asthma. Am J Respir Crit Care Med. 2016 Dec 15;194(12):1465-1474. doi: 10.1164/rccm.201602-0250OC. PMID 27367781
- [Derived] McGeachie MJ, Yates KP, Zhou X, Guo F, Sternberg AL, Van Natta ML, Wise RA, Szefler SJ, Sharma S, Kho AT, Cho MH, Croteau-Chonka DC, Castaldi PJ, Jain G, Sanyal A, Zhan Y, Lajoie BR, Dekker J, Stamatoyannopoulos J, Covar RA, Zeiger RS, Adkinson NF, Williams PV, Kelly HW, Grasemann H, Vonk JM, Koppelman GH, Postma DS, Raby BA, Houston I, Lu Q, Fuhlbrigge AL, Tantisira KG, Silverman EK, Tonascia J, Weiss ST, Strunk RC. Patterns of Growth and Decline in Lung Function in Persistent Childhood Asthma. N Engl J Med. 2016 May 12;374(19):1842-1852. doi: 10.1056/NEJMoa1513737. PMID 27168434
- [Derived] Strunk RC, Colvin R, Bacharier LB, Fuhlbrigge A, Forno E, Arbelaez AM, Tantisira KG; Childhood Asthma Management Program Research Group. Airway Obstruction Worsens in Young Adults with Asthma Who Become Obese. J Allergy Clin Immunol Pract. 2015 Sep-Oct;3(5):765-71.e2. doi: 10.1016/j.jaip.2015.05.009. Epub 2015 Jul 9. PMID 26164807
- [Derived] Drye LT, Casper AS, Sternberg AL, Holbrook JT, Jenkins G, Meinert CL. The transitioning from trials to extended follow-up studies. Clin Trials. 2014 Dec;11(6):635-47. doi: 10.1177/1740774514547396. Epub 2014 Aug 12. PMID 25115882
- [Derived] Kelly HW, Sternberg AL, Lescher R, Fuhlbrigge AL, Williams P, Zeiger RS, Raissy HH, Van Natta ML, Tonascia J, Strunk RC; CAMP Research Group. Effect of inhaled glucocorticoids in childhood on adult height. N Engl J Med. 2012 Sep 6;367(10):904-12. doi: 10.1056/NEJMoa1203229. Epub 2012 Sep 3. PMID 22938716
- [Derived] Tantisira KG, Lasky-Su J, Harada M, Murphy A, Litonjua AA, Himes BE, Lange C, Lazarus R, Sylvia J, Klanderman B, Duan QL, Qiu W, Hirota T, Martinez FD, Mauger D, Sorkness C, Szefler S, Lazarus SC, Lemanske RF Jr, Peters SP, Lima JJ, Nakamura Y, Tamari M, Weiss ST. Genomewide association between GLCCI1 and response to glucocorticoid therapy in asthma. N Engl J Med. 2011 Sep 29;365(13):1173-83. doi: 10.1056/NEJMoa0911353. Epub 2011 Sep 26. PMID 21991891
- [Derived] Hunninghake GM, Cho MH, Tesfaigzi Y, Soto-Quiros ME, Avila L, Lasky-Su J, Stidley C, Melen E, Soderhall C, Hallberg J, Kull I, Kere J, Svartengren M, Pershagen G, Wickman M, Lange C, Demeo DL, Hersh CP, Klanderman BJ, Raby BA, Sparrow D, Shapiro SD, Silverman EK, Litonjua AA, Weiss ST, Celedon JC. MMP12, lung function, and COPD in high-risk populations. N Engl J Med. 2009 Dec 31;361(27):2599-608. doi: 10.1056/NEJMoa0904006. Epub 2009 Dec 16. PMID 20018959

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between December 1993 and September 1995, 1041 children from 5 through 12 years of age with mild to moderate asthma at eight clinical centers (two HMOs associated with academic or research institutions and six located in specialty practices within academic or research institutions) were enrolled.
Pre-assignment Details: Patients were required to stop all asthma medications except as needed albuterol (prednisone could be used for asthma exacerbations) at the close of the second screening visit. Also at this time, patients began keeping a daily diary of asthma signs and symptoms, medications, school absences, and physician contacts.
Period: Overall Study
Arm/Group | 1 Budesonide | 2 Nedocromil | 3 Placebo
Started | 311 | 312 | 418
Completed | 311 | 312 | 418
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Budesonide | 2 Nedocromil | 3 Placebo | Total
Number analyzed (Participants) | 311 | 312 | 418 | 1041
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 311 | 312 | 418 | 1041
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.0 (2.1) | 8.8 (2.1) | 9.0 (2.2) | 8.9 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 106 | 184 | 420
  Male | 181 | 206 | 234 | 621
Region of Enrollment [Number; unit: participants]
  United States | 274 | 274 | 368 | 916
  Canada | 37 | 38 | 50 | 125

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Function as Measured by Normalized FEV1 Over a 4-6 Year Period
Description: Change in FEV1 % of predicted, post-bronchodilator use, from baseline to the end of treatment (4-6 years after randomization). Percent predicted determined from three separate published sets of reference equations for white, black, and Hispanic children - see NEJM 343: 1054-1062, 2000 for more details and references.
Time Frame: At the end of treatment, 4-6 years from baseline assessment
Measure: Mean (Standard Deviation); unit: percentage of predicted value
Arm/Group | 1 Budesonide | 2 Nedocromil | 3 Placebo
Number analyzed (Participants) | 306 | 307 | 411
percentage of predicted value | 0.6 (9.6) | -0.5 (9.6) | -0.1 (9.6)

2. Secondary Outcome: Bronchial Responsiveness to Serial Methacholine Concentrations Inhaled Into the Lungs
Description: Bronchial responsiveness to serial concentrations of inhaled methacholine solution (mg/ml) as measured by serial ratios of follow-up to baseline FEV1 (forced volume of air expired from the lungs in one second). A dose-response curve is calculated from the serial ratios in relation to the serial concentrations to determine PC20, the concentration associated with a 20% drop from baseline in FEV1; this PC20 is the outcome measure with units mg/ml of methacholine.
Time Frame: 4-6 years from baseline
Measure: Geometric Mean (Standard Deviation); unit: mg/ml of methacholine
Arm/Group | 1 Budesonide | 2 Nedocromil | 3 Placebo
Number analyzed (Participants) | 304 | 305 | 409
mg/ml of methacholine | 3.0 (3.3) | 1.8 (3.3) | 1.9 (3.3)

3. Secondary Outcome: Change From Baseline in the Rate of Asthma Free Days
Description: Change from baseline proportion of days without asthma symptoms or other asthma related events to proportion of days during the 4-6 years of follow-up. Asthma free days were determined from daily asthma diaries kept from baseline to the end of treatment, 4-6 years later.
Time Frame: 4-6 years from baseline
Measure: Mean (Standard Deviation); unit: days per month
Arm/Group | 1 Budesonide | 2 Nedocromil | 3 Placebo
Number analyzed (Participants) | 311 | 312 | 418
days per month | 11.3 (10.2) | 9.3 (10.2) | 9.3 (10.2)

4. Secondary Outcome: Need for Urgent Care for Asthma
Description: Counts during the period of treatment (4-6 years) of visits to emergency rooms or equivalent urgent care settings for asthma treatment.
Time Frame: 4-6 years from baseline
Measure: Number; unit: rate per 100 person years
Arm/Group | 1 Budesonide | 2 Nedocromil | 3 Placebo
Number analyzed (Participants) | 311 | 312 | 418
rate per 100 person years | 12 | 16 | 22

5. Secondary Outcome: Mortality
Description: Counts of deaths from asthma.
Time Frame: 4-6 years from baseline
Measure: Number; unit: participants
Arm/Group | 1 Budesonide | 2 Nedocromil | 3 Placebo
Number analyzed (Participants) | 311 | 312 | 418
participants | 0 | 1 | 0

6. Secondary Outcome: Change in Height From Baseline to End of Treatment, 4-6 Years Later
Description: Change in standing height from baseline to end of treatment. Standing height is measured three times without shoes using a calibrated Harpenden stadiometer; the average of the three repeated heights to the nearest 0.1 cm is the height measure at either baseline or end of treatment.
Time Frame: 4-6 years from baseline
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | 1 Budesonide | 2 Nedocromil | 3 Placebo
Number analyzed (Participants) | 311 | 312 | 418
cm | 22.7 (5.4) | 23.7 (5.4) | 23.8 (5.4)

7. Secondary Outcome: Standardized Depression Scale -- Children's Depression Inventory
Description: Change in total score on the Children's Depression Inventory from baseline to the end of treatment, 4-6 years later. The total score ranges from 0-54 with higher scores indicating greater levels of depression.
Time Frame: 4-6 years from baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 Budesonide | 2 Nedocromil | 3 Placebo
Number analyzed (Participants) | 311 | 312 | 418
units on a scale | -3.2 (5.1) | -1.8 (5.1) | -2.2 (5.1)

ADVERSE EVENTS:
Arm/Group | 1 Budesonide | 2 Nedocromil | 3 Placebo
Serious Adverse Events (participants affected / at risk) | 0/311 | 1/312 | 4/418
Other Adverse Events (participants affected / at risk) | 1/311 | 8/312 | 2/418
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Budesonide (N=311) | 2 Nedocromil (N=312) | 3 Placebo (N=418)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Psychiatric (hallucinations) (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Renal stone (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Budesonide (N=311) | 2 Nedocromil (N=312) | 3 Placebo (N=418)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal (low bone mineral density, back pain) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Phsychiatric (behavior) (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory (cough, wheeze, chest tightness, croup) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No